CLINICAL TRIAL: NCT03989206
Title: A Prospective, Multicenter, Long-Term Study to Assess the Safety and Efficacy of Nemolizumab (CD14152) in Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Long-term Safety and Efficacy of Nemolizumab With Moderate-to-severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.118163
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Moderate-to-Severe Atopic Dermatitis
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nemolizumab (Experimental): Nemolizumab administered via subcutaneous injection
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Nemolizumab — Nemolizumab
  Other Names: CD14152

SUMMARY:
Long-Term Safety and Efficacy of Nemolizumab in Subjects with Moderate-to-Severe Atopic Dermatitis Description

DETAILED DESCRIPTION:
Long-term study to assess the safety and efficacy of nemolizumab in subjects with moderate-to-severe AD

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects who may benefit from study participation in the opinion of the investigator and had participated in a prior nemolizumab study for AD
2. Female subjects of childbearing potential (ie, fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree either to be strictly abstinent throughout the study and for 12 weeks after the last study drug injection, or to use an effective and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.

Key Exclusion Criteria:

1. Subjects who, during their participation in a prior nemolizumab study, experienced an AE which in the opinion of the investigator could indicate that continued treatment with nemolizumab may present an unreasonable risk for the subject.
2. Pregnant women, breastfeeding women, or women planning a pregnancy during the clinical study.
3. Body weight < 30 kg
4. Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 2 weeks before the baseline visit, or any confirmed or suspected coronavirus disease (COVID)-19 infection within 2 weeks before the screening or baseline visit. Subjects may be rescreened once the infection has resolved. Resolution of COVID-19 infection can be confirmed by recovery assessment methods.
5. History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody)
6. Any clinically significant issue, based investigator judgement

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of TEAEs | Baseline to Week 200
Incidence of Serious TEAEs | Baseline to Week 200
Incidence and Severity of Adverse Events of Special Interest (AESIs) Throughout the Study | Baseline to Week 200

SECONDARY OUTCOMES:
Proportion of Participants with IGA score = 0-1 at Each Visit | Baseline to Week 200
Proportion of Participants with EASI-75 at Each Visit | Baseline to Week 200
Change and Percent Change From Baseline in Overall Eczema Area and Severity Index (EASI) Score at Each Visit | Baseline to Week 200
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Proportion of Participants with IGA ≤ 2 at Each Visit | Baseline to Week 200
Change and Percent Change From Baseline in SCORAD Score at Each Visit | Baseline to Week 200
Change and Percent Change From Baseline in Participant-Reported Pruritus Using 10-cm VAS (SCORAD Sub-Component) | Baseline to Week 200
Change and Percent Change From Baseline in Participant-Reported Sleep Loss Using 10-cm VAS (SCORAD Sub-Component) | Baseline to Week 200
Proportion of Participants Reporting Low Disease Activity State Based on PGAD at Each Visit | Baseline to Week 200
Proportion of Participants Satisfied with Study Treatment Based on PGAT at each visit | Baseline to Week 200
Change from Baseline in Dermatology Life Quality Index (DLQI) | Baseline to Week 200
Change From Baseline in Children's Dermatology Life Quality Index (cDLQI) Total Score at Each Visit Through Week 200 | Baseline to Week 200
Change From Baseline in Patient-Oriented Eczema Measure (POEM) Total Score at Each Visit Through Week 200 | Baseline to Week 200
Change From Baseline in Hospital Anxiety and Depression Scale (HADS) for Each Subscale at Each Visit Through Week 200 | Baseline to Week 200
Change From Baseline in Work Productivity and Activity Impairment: Atopic Dermatitis (WPAI:AD) for Each Subscale at Each Visit Through Week 200 | Baseline to Week 200
Change From Baseline in EuroQoL 5-Dimension (EQ-5D) at Each Visit Through Week 200 | Baseline to Week 200
Proportion of Participants Receiving Any Rescue Therapy by Rescue Treatment Type at Any Visit During the Treatment Period | Baseline to Week 200
Time to First Relapse | Baseline to Week 200
Duration of Remission | Baseline to Week 200
Time to Permanent Study Drug Discontinuation | Baseline to Week 200

CONTACTS AND LOCATIONS:
Locations (343):
- United States (136):
  - Galderma Investigational Site 8749, Birmingham, Alabama
  - Galderma Investigational Site 8893, Birmingham, Alabama
  - Galderma Investigational Site 8866, Guntersville, Alabama
  - Galderma Investigational Site 8808, Scottsdale, Arizona
  - Galderma Investigational Site 8873, Scottsdale, Arizona
  - Galderma Investigational Site 8447, Fort Smith, Arkansas
  - Galderma Investigational Site 8880, North Little Rock, Arkansas
  - Galderma Investigational Site 8831, Anaheim, California
  - Galderma Investigational Site 8906, Bell Gardens, California
  - Galderma Investigational Site 8456, Beverly Hills, California
  - Galderma Investigational Site 8578, Cerritos, California
  - Galderma Investigational Site 8577, Encinitas, California
  - Galderma Investigational Site 8636, Fountain Valley, California
  - Galderma Investigational Site 8224, Fremont, California
  - Galderma Investigational Site 8791, Fresno, California
  - Galderma Investigational Site 8888, Fullerton, California
  - Galderma Investigational Site 8845, Huntington Beach, California
  - Galderma Investigational Site 8833, Inglewood, California
  - Galderma Investigational Site 8686, Lomita, California
  - Galderma Investigational Site 8674, Los Angeles, California
  - Galderma Investigational Site 8683, Los Angeles, California
  - Galderma Investigational Site 8813, Los Angeles, California
  - Galderma Investigational Site 8907, Newport Beach, California
  - Galderma Investigational Site 8799, Ontario, California
  - Galderma Investigational Site 8745, Pasadena, California
  - Galderma Investigational Site 8671, San Diego, California
  - Galderma Investigational Site 8692, San Diego, California
  - Galderma Investigational Site 8658, San Diego, California
  - Galderma Investigational Site 8125, San Francisco, California
  - Galderma Investigational Site 8536, Santa Ana, California
  - Galderma Investigational Site 8608, Santa Monica, California
  - Galderma Investigational Site 8820, Westminster, California
  - Galderma Investigational Site 8637, Farmington, Connecticut
  - Galderma Investigational Site 8870, Boca Raton, Florida
  - Galderma Investigational Site 8805, Cape Coral, Florida
  - Galderma Investigational Site 8786, Clearwater, Florida
  - Galderma Investigational Site 8902, Doral, Florida
  - Galderma Investigational Site 8391, Hialeah, Florida
  - Galderma Investigational Site 8804, Hialeah, Florida
  - Galderma Investigational Site 8711, Jacksonville, Florida
  - Galderma Investigational Site 8836, Jacksonville, Florida
  - Galderma Investigational Site 8523, Largo, Florida
  - Galderma Investigational Site 8850, Margate, Florida
  - Galderma Investigational Site 8719, Miami, Florida
  - Galderma Investigational Site 8851, Miami, Florida
  - Galderma Investigational Site 8656, Miami, Florida
  - Galderma Investigational Site 8801, Miami, Florida
  - Galderma Investigational Site 8704, Miami, Florida
  - Galderma Investigational Site 8737, Miami, Florida
  - Galderma Investigational Site 8706, Miami, Florida
  - Galderma Investigational Site 8708, Miami, Florida
  - Galderma Investigational Site 8806, Miami Lakes, Florida
  - Galderma Investigational Site 8800, Miami Lakes, Florida
  - Galderma Investigational Site 8856, Ormond Beach, Florida
  - Galderma Investigational Site 8734, Pembroke Pines, Florida
  - Galderma Investigational Site 8203, Tampa, Florida
  - Galderma Investigational Site 8816, Tampa, Florida
  - Galderma Investigational Site 8889, Tampa, Florida
  - Galderma Investigational Site 8839, Tampa, Florida
  - Galderma Investigational Site 8126, West Palm Beach, Florida
  - Galderma Investigational Site 8667, Columbus, Georgia
  - Galderma Investigational Site 8744, Macon, Georgia
  - Galderma Investigational Site 8728, Newnan, Georgia
  - Galderma Investigational Site 8707, Stockbridge, Georgia
  - Galderma Investigational Site 8819, Nampa, Idaho
  - Galderma Investigational Site 9916, Chicago, Illinois
  - Galderma Investigational Site 8739, Normal, Illinois
  - Galderma Investigational Site 8729, Rolling Meadows, Illinois
  - Galderma Investigational Sites 8571, Skokie, Illinois
  - Galderma Investigational Site 8712, Skokie, Illinois
  - Galderma Investigational Site 8142, Indianapolis, Indiana
  - Galderma Investigational Site 8724, New Albany, Indiana
  - Galderma Investigational Site 9934, Shawnee Mission, Kansas
  - Galderma Investigational Site 8771, Louisville, Kentucky
  - Galderma Investigational Site 8882, Bangor, Maine
  - Galderma Investigational Site 8743, Ann Arbor, Michigan
  - Galderma Investigational Site 8512, Bay City, Michigan
  - Galderma Investigational Site 8554, Detroit, Michigan
  - Galderma Investigational Site 8617, Farmington Hills, Michigan
  - Galderma Investigational Site 8155, Troy, Michigan
  - Galderma Investigational Site 8849, Troy, Michigan
  - Galderma Investigational Site 8226, Warren, Michigan
  - Galderma Investigational Site 8748, Ypsilanti, Michigan
  - Galderma Investigational Site 8521, Saint Joseph, Missouri
  - Galderma Investigational Site 8718, Missoula, Montana
  - Galderma Investigational Site 8810, Omaha, Nebraska
  - Galderma Investigational Site 8740, Henderson, Nevada
  - Galderma Investigational Site 8825, Las Vegas, Nevada
  - Galderma Investigational Site 8675, Las Vegas, Nevada
  - Galderma Investigational Site 8109, Lebanon, New Hampshire
  - Galderma Investigational Site 8506, Hackensack, New Jersey
  - Galderma Investigational Site 8826, Albuquerque, New Mexico
  - Galderma Investigational Site 8242, Brooklyn, New York
  - Galderma Investigational Site 8741, Buffalo, New York
  - Galderma Investigational Site 8723, Cortland, New York
  - Galderma Investigational Site 8828, Forest Hills, New York
  - Galderma Investigational Site 9925, Glendale, New York
  - Galderma Investigational Site 8733, New York, New York
  - Galderma Investigational Site 8620, New York, New York
  - Galderma Investigational Site 8279, New York, New York
  - Galderma Investigational Site 8772, Durham, North Carolina
  - Galderma Investigational Site 8795, Shelby, North Carolina
  - Galderma Investigational Site 8726, Wilmington, North Carolina
  - Galderma Investigational Site 8648, Wilmington, North Carolina
  - Galderma Investigational Site 8702, Bexley, Ohio
  - Galderma Investigational Site 8747, Cincinnati, Ohio
  - Galderma Investigational Site 8595, Dublin, Ohio
  - Galderma Investigational Site 8206, Norman, Oklahoma
  - Galderma Investigational Site 8857, Oklahoma City, Oklahoma
  - Galderma Investigational Site 8212, Portland, Oregon
  - Galderma Investigational Site 8255, Philadelphia, Pennsylvania
  - Galderma Investigational Site 8721, Pittsburgh, Pennsylvania
  - Galderma Investigational Site 8802, Plymouth Meeting, Pennsylvania
  - Galderma Investigational Site 8777, Charleston, South Carolina
  - Galderma Investigational Site 8736, Charleston, South Carolina
  - Galderma Investigational Site 8713, North Charleston, South Carolina
  - Galderma Investigational Site 8818, Rapid City, South Dakota
  - Galderma Investigational Site 8133, Arlington, Texas
  - Galderma Investigational Site 8298, Austin, Texas
  - Galderma Investigational Site 8238, Dallas, Texas
  - Galderma Investigational Site 8245, Dallas, Texas
  - Galderma Investigational Site 8827, Dripping Springs, Texas
  - Galderma Investigational Site 8664, Frisco, Texas
  - Galderma Investigational Site 8807, Houston, Texas
  - Galderma Investigational Site 8042, Houston, Texas
  - Galderma Investigational Site 8670, Houston, Texas
  - Galderma Investigational Site 8817, Katy, Texas
  - Galderma Investigational Site 8787, Plano, Texas
  - Galderma Investigational Site 8329, San Antonio, Texas
  - Galderma Investigational Site 8618, Waco, Texas
  - Galderma Investigational Site 8003, Webster, Texas
  - Galderma Investigational Site 8672, Salt Lake City, Utah
  - Galderma Investigational Site 8738, Burke, Virginia
  - Galderma Investigational Site 8862, Fairfax, Virginia
  - Galderma Investigational Site 8896, Richmond, Virginia
  - Galderma Investigational Site 8434, Seattle, Washington
- Australia (11):
  - Galderma Investigational Site 5441, Darlinghurst, New South Wales
  - Galderma Investigational Site 5759, Kogarah, New South Wales
  - Galderma Investigational Site 6152, Westmead, New South Wales
  - Galderma Investigational Site 5638, Benowa, Queensland
  - Galderma Investigational Site 6161, Brisbane, Queensland
  - Galderma Investigational Site 6159, Woodville, South Australia
  - Galderma Investigational Site 6131, Carlton, Victoria
  - Galderma Investigational Site 5366, East Melbourne, Victoria
  - Galderma Investigational Site 5458, Parkville, Victoria
  - Galderma Investigational Site 6160, Parkville, Victoria
  - Galderma Investigational Site 6153, Victoria Park, Western Australia
- Austria (4):
  - Galderma Investigational Site 6157, Graz, Styria
  - Galderma Investigational Site 6156, Linz, Upper Austria
  - Galderma Investigational Site 6194, Vienna
  - Galderma Investigational Site 6158, Vienna
- Belgium (5):
  - Galderma Investigational Site 6038, Leuven, Vlaams-Brabant
  - Galderma Investigational Site 5448, Brussels
  - Galderma Investigational Site 6163, Edegem
  - Galderma Investigational Site 6164, Ghent
  - Galderma Investigational Site 6162, Liège
- Bulgaria (13):
  - Galderma Investigational Site 6029, Pleven
  - Galderma Investigational Site 6051, Sofia
  - Galderma Investigational Site 6078, Sofia
  - Galderma Investigational Site 6102, Sofia
  - Galderma Investigational Site 6165, Sofia
  - Galderma Investigational Site 6216, Sofia
  - Galderma Investigational Site 6046, Sofia
  - Galderma Investigational Site 6080, Sofia
  - Galderma Investigational Site 6101, Sofia
  - Galderma Investigational Site 6079, Sofia
  - Galderma Investigational Site 6250, Sofia
  - Galderma Investigational Site 6136, Stara Zagora
  - Galderma Investigational Site 6251, Stara Zagora
- Canada (15):
  - Galderma Investigational Site 8085, Calgary, Alberta
  - Galderma Investigational Site 8903, Calgary, Alberta
  - Galderma Investigational Site 8215, Calgary, Alberta
  - Galderma Investigational Site 8824, Edmonton, Alberta
  - Galderma Investigational Site 8722, Edmonton, Alberta
  - Galderma Investigational Site 8161, Surrey, British Columbia
  - Galderma Investigational Site 8586, Barrie, Ontario
  - Galderma Investigational Site 8904, Guelph, Ontario
  - Galderma Investigational Site 8780, Niagara Falls, Ontario
  - Galderma Investigational Site 8610, Ottawa, Ontario
  - Galderma Investigational Site 8901, Ottawa, Ontario
  - Galderma Investigational Site 8336, Toronto, Ontario
  - Galderma Investigational Site 8899, Toronto, Ontario
  - Galderma Investigational Site 8731, Waterloo, Ontario
  - Galderma Investigational Site 8000, Saint John
- Czechia (8):
  - Galderma Investigational Site 6055, Brno
  - Galderma Investigational Site 5225, Náchod
  - Galderma Investigational Site 6030, Olomouc
  - Galderma Investigational Site 6024, Prague
  - Galderma Investigational Site 6021, Prague
  - Galderma Investigational Site 6054, Prague
  - Galderma Investigational Site 6240, Prague
  - Galderma Investigational Site 6025, Prague
- Estonia (3):
  - Galderma Investigational Site 6068, Tallinn
  - Galderma Investigational Site 6069, Tallinn
  - Galderma Investigational Site 6067, Tartu
- France (12):
  - Galderma Investigational Site 6198, Le Mans
  - Galderma Investigational Site 5031, Lille
  - Galderma Investigational Site 6170, Martigues
  - Galderma Investigational Site 6167, Nantes
  - Galderma Investigational Site 5140, Nice
  - Galderma Investigational Site 6133, Paris
  - Galderma Investigational Site 6166, Paris
  - Galderma Investigational Site 5407, Pierre-Bénite
  - Galderma Investigational Site 6135, Quimper
  - Galderma Investigational Site 6197, Toulon
  - Galderma Investigational Site 6169, Toulouse
  - Galderma Investigational Site 6168, Valence
- Georgia (8):
  - Galderma Investigational Site 6224, Tbilisi
  - Galderma Investigational Site 6228, Tbilisi
  - Galderma Investigational Site 6235, Tbilisi
  - Galderma Investigational Site 6238, Tbilisi
  - Galderma Investigational Site 6227, Tbilisi
  - Galderma Investigational Site 6230, Tbilisi
  - Galderma Investigational Site 6234, Tbilisi
  - Galderma Investigational Site 6236, Zugdidi
- Germany (26):
  - Galderma Investigational Site 5482, Aachen
  - Galderma Investigational Site 5566, Augsburg
  - Galderma Investigational Site 6022, Bad Bentheim
  - Galderma Investigational Site 6110, Berlin
  - Galderma Investigational Site 6061, Bielefeld
  - Galderma Investigational Site 6082, Bonn
  - Galderma Investigational Site 6062, Buxtehude
  - Galderma Investigational Site 5368, Darmstadt
  - Galderma Investigational Site 6132, Dresden
  - Galderma Investigational Site 6028, Dülmen
  - Galderma Investigational Site 6031, Düsseldorf
  - Galderma Investigational Site 5442, Gera
  - Galderma Investigational Site 6081, Goettigen
  - Galderma Investigational Site 6062, Halle
  - Galderma Investigational Site 6041, Hamburg
  - Galderma Investigational Site 6150, Hamburg
  - Galderma Investigational Site 6040, Hamburg
  - Galderma Investigational Site 5469, Heidelberg
  - Galderma Investigational Site 6086, Kiel
  - Galderma Investigational Site 6146, Langenau
  - Galderma Investigational Site 6084, Mainz
  - Galderma Investigational Site 5382, Munich
  - Galderma Investigational Site 6039, Münster
  - Galderma Investigational Site 5918, Osnabrück
  - Galderma Investigational Site 6109, Stuttgart
  - Galderma Investigational Site 6214, Tübingen
- Hungary (6):
  - Galderma Investigational Site 6147, Budapest
  - Galderma Investigational Site 5513, Budapest
  - Galderma Investigational Site 5567, Debrecen
  - Galderma Investigational Site 6026, Debrecen
  - Galderma Investigational Site 6254, Gyula
  - Galderma Investigational Site 6053, Veszprém
- Italy (6):
  - Galderma Investigational Site 6145, Bologna
  - Galderma Investigational Site 6045, L’Aquila
  - Galderma Investigational Site 6049, Roma
  - Galderma Investigational Site 6177, Rome
  - Galderma Investigational Site 6155, Rozzano
  - Galderma Investigational Site 6175, Vicenza
- Latvia (4):
  - Galderma Investigational Site 6113, Liepāja
  - Galderma Investigational Site 6134, Riga
  - Galderma Investigational Site 6059, Riga
  - Galderma Investigational Site 6060, Talsi
- Lithuania (3):
  - Galderma Investigational Site 6111, Kaunas
  - Galderma Investigational Site 6073, Vilnius
  - Galderma Investigational Site 6112, Vilnius
- Netherlands (3):
  - Galderma Investigational Site 6212, Groningen
  - Galderma Investigational Site 6108, Rotterdam
  - Galderma Investigational Site 6027, Utrecht
- New Zealand (2):
  - Galderma Investigational Site 6119, Hamilton
  - Galderma Investigational Site 6118, Wellington
- Poland (38):
  - Galderma Investigational Site 5773, Bialystok
  - Galderma Investigational Site 6097, Chorzów
  - Galderma Investigational Site 6255, Częstochowa
  - Galderma Investigational Site 6075, Gdansk
  - Galderma Investigational Site 6243, Gdansk
  - Galderma Investigational Site 5138, Gdansk
  - Galderma Investigational Site 6244, Gdynia
  - Galderma Investigational Site 6087, Katowice
  - Galderma Investigational Site 5021, Katowice
  - Galderma Investigational Site 5362, Krakow
  - Galderma Investigational Site 6052, Krakow
  - Galderma Investigational Site 6245, Lodz
  - Galderma Investigational Site 5570, Lodz
  - Galderma Investigational Site 5363, Lodz
  - Galderma Investigational Site 6231, Lodz
  - Galderma Investigational Site 5367, Lublin
  - Galderma Investigational Site 6071, Lublin
  - Galderma Investigational Site 5377, Nowa Sól
  - Galderma Investigational Site 6063, Olsztyn
  - Galderma Investigational Site 6237, Ostrowiec Świętokrzyski
  - Galderma Investigational Site 6085, Poznan
  - Galderma Investigational Site 6127, Poznan
  - Galderma Investigational Site 5495, Rzeszów
  - Galderma Investigational Site 6088, Rzeszów
  - Galderma Investigational Site 6223, Szczecin
  - Galderma Investigational Site 6130, Szczecin
  - Galderma Investigational Site 6048, Tarnów
  - Galderma Investigational Site 6126, Warsaw
  - Galderma Investigational Site 6065, Warsaw
  - Galderma Investigational Site 5707, Warsaw
  - Galderma Investigational Site 6122, Warsaw
  - Galderma Investigational Site 6242, Warsaw
  - Galderma Investigational Site 6064, Warsaw
  - Galderma Investigational Site 6222, Warsaw
  - Galderma Investigational Site 6047, Wroclaw
  - Galderma Investigational Site 6185, Wroclaw
  - Galderma Investigational Site 6096, Wroclaw
  - Galderma Investigational Site 5005, Wroclaw
- Singapore (3):
  - Galderma Investigational Site 6124, Singapore
  - Galderma Investigational Site 6077, Singapore
  - Galderma Investigational Site 5499, Singapore
- South Korea (15):
  - Galderma Investigational Site 6095, Bucheon-si
  - Galderma Investigational Site 6100, Busan
  - Galderma Investigational Site 6098, Gyeonggi-do
  - Galderma Investigational Site 6154, Gyeonggi-do
  - Galderma Investigational Site 6138, Incheon
  - Galderma Investigational Site 6120, Incheon
  - Galderma Investigational Site 6093, Incheon
  - Galderma Investigational Site 6105, Seoul
  - Galderma Investigational Site 5659, Seoul
  - Galderma Investigational Site 6116, Seoul
  - Galderma Investigational Site 6129, Seoul
  - Galderma Investigational Site 6103, Seoul
  - Galderma Investigational Site 6056, Seoul
  - Galderma Investigational Site 6094, Seoul
  - Galderma Investigational Site 6099, Seoul
- Spain (12):
  - Galderma Investigational Site 6057, Alicante
  - Galderma Investigational Site 6037, Barcelona
  - Galderma Investigational Site 6035, Barcelona
  - Galderma Investigational Site 5580, L'Hospitalet de Llobregat
  - Galderma Investigational Site 6106, Las Palmas de Gran Canaria
  - Galderma Investigational Site 6058, Madrid
  - Galderma Investigational Site 5842, Madrid
  - Galderma Investigational Site 6190, Madrid
  - Galderma Investigational Site 6186, Madrid
  - Galderma Investigational Site 6036, Madrid
  - Galderma Investigational Site 5551, Madrid
  - Galderma Investigational Site 6191, Pamplona
- United Kingdom (10):
  - Galderma Investigational Site 6202, Barnsley
  - Galderma Investigational Site 6207, Blackpool
  - Galderma Investigational Site 6203, Cannock
  - Galderma Investigational Site 6090, Dudley
  - Galderma Investigational Site 6104, Glasgow
  - Galderma Investigational Site 6204, Liverpool
  - Galderma Investigational Site 6121, London
  - Galderma Investigational Site 6205, Manchester
  - Galderma Investigational Site 6208, Newcastle
  - Galderma Investigational Site 6206, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augustin M, Tauber M, Sidbury R, Silverberg JI, Papp KA, Thaci D, De Bruin-Weller MS, Reich A, Peris K, Barber K, Galus R, Kaszuba A, Zirwas M, Nahm WK, Trullenque G, Maintz L, Alpizar S, Son SW, Laquer V, Gold LS, Cheong SY, Ryzhkova A, Drahos A, Ulianov L, Piketty C. Safety and efficacy of nemolizumab for atopic dermatitis up to 2 years in open-label extension study. J Eur Acad Dermatol Venereol. 2025 Oct 13. doi: 10.1111/jdv.70080. Online ahead of print. PMID 41081535
- [Derived] Brunner PM. A novel treatment approach for atopic dermatitis. Lancet. 2024 Aug 3;404(10451):407-409. doi: 10.1016/S0140-6736(24)01488-0. Epub 2024 Jul 25. No abstract available. PMID 39068954